CLINICAL TRIAL: NCT01208922
Title: A Randomised, Double-blind, Double-dummy, Multi-centre, Comparative Parallel-group Study to Evaluate the Efficacy and Safety of Oral Daily Rifamycin SV-MMX® 400 mg b.i.d. vs. Ciprofloxacin 500 mg b.i.d. in the Treatment of Acute Infectious Diarrhoea in Travellers
Brief Title: Rifamycin SV-MMX® Tablets Versus Ciprofloxacin Capsules in Acute Traveller's Diarrhoea
Acronym: ERASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIT-1/AID
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-10

CONDITIONS: Traveler's Diarrhea
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Rifamycin SV-MMX® 200 mg tablets
  Interventions: Drug: Rifamycin SV-MMX®
- Group B (Active Comparator): Ciprofloxacin 500 mg capsules
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Rifamycin SV-MMX® — 2 Rifamycin SV-MMX® 200 mg tablets and 1 placebo to ciprofloxacin capsule, b.i.d.
  Arms: Group A
Drug: Ciprofloxacin — 1 ciprofloxacin 500 mg capsule and 2 placebos to Rifamycin SV-MMX® 200 mg tablets, b.i.d.
  Arms: Group B

SUMMARY:
The purpose of this study is to prove the non-inferiority of Rifamycin SV-MMX® versus Ciprofloxacin for the treatment of adults with traveller's diarrhoea.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Men or women between 18 and 85 years of age,
* History of arriving from their country of residence in the industrialized part of the world within the past 4 weeks,
* Presenting with acute infectious diarrhoea (defined as at least 3 unformed, watery or soft stools accompanied by symptoms within 24 hours preceding randomisation with duration of illness ≤ 72 hours),
* Presence of one or more signs or symptoms of enteric infection (moderate to severe gas/flatulence, nausea, vomiting, abdominal cramps or pain, rectal tenesmus, fecal urgency),
* Women of childbearing potential had to apply during the entire duration of the study a highly effective method of birth control

Exclusion Criteria:

* Residency in any country with high incidence rate of TD within the past 6 months,
* Fever (defined as a body (oral) temperature >100.4°F or 38.0°C; antipyretic medication should not have been administered in the 6 hours prior to this assessment),
* Known or suspected infection with non-bacterial pathogen,
* Presence of diarrhoea of >72 hours duration,
* Presence of grossly bloody stool,
* Presence of moderate or severe dehydration (i.e. symptoms of hypovolemia such as orthostatic hypotension, dizziness or wrinkling of skin),
* History of inflammatory bowel disease or celiac disease,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Robert Steffen, M. D., Principal Investigator — University of Zurich, Switzerland
Locations (19):
- Site 401, Quito, Ecuador
- Site 200, Quetzaltenango, Guatemala
- India (17):
  - Site 101, Mapusa, Karaswada
  - Site 124, Ajmer
  - Site 118, Bardez
  - Site 120, Calangute
  - Site 104, Hyderabad
  - Site 114, Kolkata
  - Site 116, Lucknow
  - Site 107, Madgaon
  - Site 110, Madgaon
  - Site 123, New Delhi
  - Site 122, Panjim
  - Site 102, Puducherry
  - Site 115, Pushkar
  - Site 119, Salcette
  - Site 111, Tiswadi
  - Site 109, Varanasi
  - Site 103, Vijayawada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from November 2010 until January 2016
Pre-assignment Details: A total of 835 patients were enrolled and were randomised to one of the 2 treatment groups according to the randomisation plan. All randomised patients received at least one dose of study medication.
Groups:
- Rifamycin Group: Rifamycin SV-MMX® 200 mg tablets
  Rifamycin SV-MMX®: 2 Rifamycin SV-MMX® 200 mg tablets and 1 placebo to ciprofloxacin capsule, b.i.d.
- Ciprofloxacin Group: Ciprofloxacin 500 mg capsules
  Ciprofloxacin: 1 ciprofloxacin 500 mg capsule and 2 placebos to Rifamycin SV-MMX® 200 mg tablets, b.i.d.
Period: Overall Study
Arm/Group | Rifamycin Group | Ciprofloxacin Group
Started | 420 | 415
Completed | 409 | 405
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Population: Baseline results were reported for Full Analysis Set, which included all randomised patients (as randomised) who received at least one dose of study medication. Patients with uncertainty as to whether they had received study medication or not (e.g., due to lost to follow-up) were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 420 | 415 | 835
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (16.1) | 40.4 (16.6) | 40.2 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 197 | 412
  Male | 205 | 218 | 423
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 75 | 68 | 143
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 342 | 344 | 686
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Ecuador | 1 | 0 | 1
  Guatemala | 14 | 15 | 29
  India | 405 | 400 | 805

OUTCOME MEASURES:

1. Primary Outcome: Time to Last Unformed Stool (TLUS)
Description: Time to Last Unformed Stool (TLUS), defined as the interval in hours between the first dose of study drug and the last unformed stool passed, after which clinical cure was declared.
Time Frame: 5 days
Population: Efficacy results were reported for Full Analysis Set, which all randomised patients (as randomised) who received at least one dose of study medication. Patients with uncertainty as to whether they had received study medication or not (e.g., due to lost to follow-up) were included.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Group A | Group B
Number analyzed (Participants) | 420 | 415
hours | 44.3 [40.1 to 47.5] | 40.3 [33.5 to 44.8]

2. Secondary Outcome: Number of Patients With Clinical Cure
Description: Clinical Cure Rate: 24-hour period with no clinical symptoms except mild flatulence, no fever, no watery stools and no more than 2 soft stools OR 48-hour period with no stools or only formed stools, and no fever, with our without symptoms of enteric infection.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 420 | 415
Participants | 357 | 352

ADVERSE EVENTS:
Time Frame: An average of 1 month
Description: Non-serious AEs were analysed as Treatment-Emergent AEs defined as all AEs with onset after treatment day 1 but not after the last day with study drug administration.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/420 | 0/415
Serious Adverse Events (participants affected / at risk) | 0/420 | 0/415
Other Adverse Events (participants affected / at risk) | 36/420 | 32/415
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=420) | Group B (N=415)
Headache (Nervous system disorders) | 13 (13) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Flatulence (Gastrointestinal disorders) | 5 (5) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No